CLINICAL TRIAL: NCT00940823
Title: The Ahmed Versus Baerveldt (AVB) Study: Prospective, Multicenter Trial Comparing the Ahmed-FP7 Valve With the Baerveldt-350 Implant in Treating Refractory Glaucoma
Brief Title: The AVB Study: Prospective Study Comparing the Ahmed Valve and the Baerveldt Implant for Treating Refractory Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Credit Valley EyeCare (Industry)
Collaborators: Glaucoma Research Society of Canada (Other)
Responsible Party: Principal Investigator, Panos G. Christakis, Study Director, Credit Valley EyeCare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVEC-AVB; GRSC-2005 (Other: Glaucoma Research Society of Canada)
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Glaucoma
Keywords: Glaucoma Drainage Device; Aqueous Shunt Implant; Ahmed Valve; Baerveldt Tube; Refractory Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ahmed FP7 Valve (Active Comparator): Ahmed valve glaucoma drainage device implant for treatment of refractory glaucoma.
  Interventions: Device: Ahmed FP7 Valve
- Baerveldt-350 Tube (Active Comparator): Baerveldt tube glaucoma drainage device implant for treatment of refractory glaucoma.
  Interventions: Device: Baerveldt-350 Tube

INTERVENTIONS:
Device: Ahmed FP7 Valve — Implantation of Ahmed FP7 Valve to lower intraocular pressure in refractory glaucoma.
  Other Names: New World Medical; AGV FP7
  Arms: Ahmed FP7 Valve
Device: Baerveldt-350 Tube — Implantation of Baerveldt-350 Tube to lower intraocular pressure in refractory glaucoma.
  Other Names: Advanced Medical Optics; BG 101-350
  Arms: Baerveldt-350 Tube

SUMMARY:
The purpose of this study is to compare the safety and efficacy of the Ahmed valve and the Baerveldt implant in treating refractory glaucoma. Eligible patients will be recruited from multiple study centers and randomized to a glaucoma drainage device for implantation. They will be followed long-term based upon outcome measures including intraocular pressure, glaucoma medication use, visual acuity, complications of the surgery and further treatments required.

DETAILED DESCRIPTION:
Introduction:

The use of a glaucoma drainage device (GDD) is indicated in cases of refractory glaucoma not responsive to conventional medication, laser and surgical therapy. Most of these patients are at high risk for surgical failure, with serious concomitant ocular and systemic diseases. GDD's are increasingly being used to obtain low target intraocular pressures (IOP) in patients who have failed antimetabolite trabeculectomy or have active neovascular glaucoma.

Since Molteno's original design, several drainage devices have become commercially available for implantation. Currently, the two most commonly used devices are the Ahmed Glaucoma Valve (AGV) (New World Medical, Inc., Rancho Cucamonga, CA), and the Baerveldt Glaucoma Device (BGD) (Advanced Medical Optics, Santa Ana, CA). The AGV, with a venture-based flow-restrictive valve is helpful in minimizing postoperative hypotony and complications associated with hypotony, including flat anterior chamber, choroidal effusions, and suprachoroidal hemorrhage. However, there appears to be a high rate of encapsulation and hypertension associated with this device, and increased requirement of postoperative glaucoma medication use. The BGD, a non-valved device, requires early ligature of flow by the use of a suture restriction to allow adequate time for bleb formation. Although this can result in an initial post-operative hypertension phase, it results in less encapsulation and theoretically fewer postoperative glaucoma medications and better IOP control. However, the lack of a flow-restrictor and the large filtering surface area may result in a greater risk for hypotony related complications.

Although several studies comparing the AGV and BGD have been reported, they have all been retrospective, nonrandomized, small scale, and compare different patient populations. The results have been inconclusive and conflicting in evaluating the relative efficacy and characteristics of these two devices, and further research needs to be done in order to answer these questions.

Objective:

The Ahmed vs. Baerveldt (AVB) Study is the first multicenter prospective randomized clinical trial comparing the Ahmed FP7 valve and the Baerveldt-350 tube shunt glaucoma drainage devices. Primary outcome is surgical failure, a composite criteria evaluating the intraocular pressure lowering effect of the devices, complications of the surgery, treatments for complications, glaucoma medication use, and the preservation of visual acuity. Secondary outcomes will evaluate these variables individually, and any non-glaucoma related ocular pathology and required interventions.

AVB Study Manual:

An AVB Study Manual including the study design and protocol, standardized surgical technique, patient education and consent form, and data collection protocol was distributed to each clinical site. The contents of the manual received ethics approval by the Institutional Review Board (IRB) at the primary site.

Study Organization:

1. Investigator Committee (IC): Composed of study investigators and under the leadership of the Study Chair. The IC's responsibilities are defined below:

   1. Designing the study protocol to ensure valid scientific method and proper ethical conduct.
   2. Overseeing clinical centers to ensure that the protocol and ethical standards of the study are being upheld.
   3. Overseeing the Data Acquisition & Statistical Center to ensure that all practices are in accordance with those outlined in the protocol, and meet the ethical standards of the study.
   4. Drafting and editing study documents critically for intellectual content and ethical considerations.
2. Clinical Centers (CC): Composed of study sites led by a Site Primary Investigator, whose responsibilities are defined below:

   1. Enrolling patients in the study after determining eligibility and providing patient education. Informed consent must be written.
   2. Ensuring that the study protocol and ethical standards of the study are upheld.
   3. Ensuring that the study adheres to the policies set forth by the local Institutional/Ethical Review Board.
   4. Acquiring study data and making it available to the Data Monitoring & Statistics Committee.
3. Data Acquisition & Statistical Center (DASC): Composed of Study Director and Study Statistician, with the following responsibilities:

   1. Acquiring study data from each Clinical Center using the online study database (http://www.avsbstudy.com)
   2. Statistical analysis of the study data.

Methods:

Patient Enrollment and Treatment Assignment:

Patients were recruited from 7 study sites by 10 surgeons. After patient eligibility and written informed consent was obtained by the Site PI, randomization to placement of an Ahmed FP7 valve or a Baerveldt-350 tube shunt was made by coin toss.

Pre-operative data collection:

The following data was collected in the 3 months prior to surgery: date of birth, gender, race, glaucoma diagnosis and etiology, past ocular history (diagnoses, surgical and laser procedures), best corrected visual acuity, intraocular pressure, glaucoma medication use, abnormal slit lamp findings, and abnormal fundus exam findings.

Surgical Procedure:

The surgical procedures used for the AVB Study are standardized, and any complications during surgery will be noted and defined.

Ahmed FP7 valve implantation:

A superior or inferior corneal traction suture with 8-0 Vicryl was placed for globe fixation as required. A 90-degree conjunctival peritomy was followed by blunt dissection to mobilize a fornix or limbus-based conjunctival flap over the area of intended device implantation. Non-preserved lidocaine 1% was injected under the conjunctival flap, posteriorly, and under the extraocular muscle bellies with a blunt cannula. Gentle cautery was used to obtain hemostasis.

The Ahmed Glaucoma Valve model FP-7 was primed with balanced salt solution, and placed in the intended quadrant. The plate was sutured to sclera 8-10mm posterior to the limbus with two 8-0 or 10-0 Nylon sutures.

A paracentesis was made if required, and a viscoelastic agent used to form the anterior chamber. A 22-gauge needle was used to create needle tract into the anterior chamber.

The tube was trimmed, and placed into the anterior chamber through the needle tract. The tube was attached to the sclera using a 10-0 Nylon suture if required. A sclera or corneal graft was placed over the tube and sutured to the sclera with 10-0 Nylon.

The conjunctival flap was closed with 8-0 or 10-0 Vicryl suture. At the conclusion of the case, Maxitrol ointment was placed on the eye. No patients were patched, although shields were given to patients. That day, patients were started on antibiotic and steroid eye drops. A cycloplegic was used as indicated.

Baerveldt-350 tube shunt implantation:

A superior or inferior corneal traction suture with 8-0 Vicryl was placed for globe fixation. A 90 to 120-degree conjunctival peritomy was followed by blunt dissection to mobilize a fornix or limbus-based conjunctival flap over the area of intended device implantation. Non-preserved lidocaine 1% was injected under the conjunctival flap, posteriorly, and under the extraocular muscle bellies with a blunt cannula. Gentle cautery was used to obtain hemostasis.

Both adjacent extraocular muscles were isolated using a muscle hook. 4-0 silk sutures were used for fixation if necessary.

The Baerveldt drainage device model BG101-350 was checked with balanced salt solution, and a 4-0 Nylon releasable intraluminal suture was placed. A 7-0 or 8-0 Vicryl ligature suture was placed around the tube. The plate was placed in the intended quadrant and under the muscle bellies. The plate was sutured to the sclera 8-12mm posterior to the limbus with two 8-0 or 10-0 Nylon sutures.

A paracentesis was made if it was required, and a viscoelastic agent used to form the anterior chamber. A 22-gauge needle was used to create needle tract into the anterior chamber. The tube was trimmed, and placed into the anterior chamber through the needle tract. The tube was attached to the sclera using a 10-0 Nylon suture if required. A sclera or corneal graft was placed over the tube and sutured to the sclera.

The conjunctival flap was closed with an 8-0 or 10-0 Vicryl suture. At the conclusion of the case, Atropine 1% drops and Maxitrol ointment was placed on the eye. No patients were patched, although shields were given to patients. On the day of surgery, patients were started on antibiotics and steroid eye drops. A cycloplegic agent was used as indicated.

Post-operative data collection:

Patients were seen post-operatively at a minimum of 1 day, 1 week, 2 weeks, 1 month, 2 months, 3 months, 6 months, 12 months, 18 months 2 years, 3 years, 4 years and 5 years. Further visits were made as deemed necessary. At each visit, the following data was collected:

1. Intraocular pressure (IOP) by Goldmann Applanation Tonometry
2. Visual Acuity (VA) using a Snellen Chart or Low Vision Chart
3. Glaucoma Medication Use
4. Slit Lamp Biomicroscopy & Ophthalmoscopy
5. Complications of Surgery
6. Interventions/Treatment of Complications

Outcome measures:

Based upon the pre-operative data and post-operative results, a study outcome will be assigned to each patient, as defined below:

Complete Success: (requires all of the following criteria)

1. IOP: 5 mmHg <= IOP <= 18 mmHg with a reduction in IOP of 20% or greater from baseline at every visit after 3 months.
2. Medications: No anti-glaucoma medications are required.
3. Complications: No vision threatening complications related to the implant/surgery.
4. Interventions: No additional glaucoma surgery or laser procedures are allowed.
5. Vision: No greater than a doubling of the mean angle of resolution (logMAR), which corresponds to approximately 2 Snellen lines.

Qualified Success: (requires all of the following criteria)

1. IOP: 5 mmHg <= IOP <= 18 mmHg with a reduction in IOP of 20% or greater from baseline, with no two consecutive visits after 3 months which do not meet this criterion.
2. Medications: Anti-glaucoma medications may be used.
3. Surgery/Complications: No vision threatening complications or surgery occurred after implantation of the GDD.
4. Interventions: Surgical and laser interventions to correct non-vision threatening complications of implant/surgery are allowed, but no additional glaucoma procedures are allowed.
5. Vision: No progression to no light perception.

Failure: (if any of the following criteria are met)

1. IOP: IOP <5 mmHg or >18 mmHg or reduction <20% from pre-operative IOP in two consecutive visits after 3 months.
2. Surgery/Complications: Vision threatening complications or surgery required that is related to the implant. This includes severe choroidal effusions requiring drainage, suprachoroidal hemorrhage, endophthalmitis or malignant glaucoma requiring surgery.
3. Interventions: An additional glaucoma procedure is required (e.g. cyclodestruction, gold shunt implantation).
4. Vision: Progression to no light perception.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18.
* Inadequately controlled glaucoma determined as intraocular pressure (IOP) greater than target, which has not responded to conventional medical and surgical therapy.
* Patients with significant conjunctival scarring or high-risk disease (active neovascular glaucoma) precluding antimetabolite trabeculectomy will be included in the study.
* Provide written informed consent to participate in the study.

Exclusion Criteria:

* Age less than 18.
* Patient will undergo an additional procedure at the time of glaucoma drainage device implantation (i.e. lensectomy, penetrating keratoplasty)
* No light perception vision.
* Patient has already been enrolled in the study in the contralateral eye.
* Patient is unwilling or unable to provide informed consent to participate in the study, or adhere to the study requirements including implant randomization and required follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2005-07; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal K Ahmed, MD, Study Chair — University of Toronto Department of Ophthalmology & Vision Sciences; Panos G Christakis, BS, Study Director — Yale University; James C Tsai, MD, Principal Investigator — Yale Ophthalmology & Visual Science; Jeffrey W Kalenak, MD, Principal Investigator — Drs. Massaro & Kalenak, SC; Louis B Cantor, MD, Principal Investigator — Department of Ophthalmology, Indiana University; Jeffrey A Kammer, MD, Principal Investigator — Department of Ophthalmology and Visual Sciences: Vanderbilt University, School of Medicine; Paul J Harasymowycz, MD, Principal Investigator — University of Montreal: Department of Ophthalmology; Juan J Mura, MD, Principal Investigator — Clinic of Las Condes
Locations (6):
- United States (3):
  - Eugene and Marilyn Glick Eye Institute, Indianapolis, Indiana
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Drs. Massaro and Kalenak, Milwaukee, Wisconsin
- Canada (2):
  - Credit ValleyEC, Toronto, Ontario
  - Montreal Glaucoma Institute, Montreal, Quebec
- Clinic of Las Condes, Santiago, Chile

REFERENCES:
- [Background] Syed HM, Law SK, Nam SH, Li G, Caprioli J, Coleman A. Baerveldt-350 implant versus Ahmed valve for refractory glaucoma: a case-controlled comparison. J Glaucoma. 2004 Feb;13(1):38-45. doi: 10.1097/00061198-200402000-00008. PMID 14704542
- [Background] Wang JC, See JL, Chew PT. Experience with the use of Baerveldt and Ahmed glaucoma drainage implants in an Asian population. Ophthalmology. 2004 Jul;111(7):1383-8. doi: 10.1016/j.ophtha.2003.11.005. PMID 15234141
- [Background] Tsai JC, Johnson CC, Dietrich MS. The Ahmed shunt versus the Baerveldt shunt for refractory glaucoma: a single-surgeon comparison of outcome. Ophthalmology. 2003 Sep;110(9):1814-21. doi: 10.1016/S0161-6420(03)00574-8. PMID 13129882
- [Background] Tsai JC, Johnson CC, Kammer JA, Dietrich MS. The Ahmed shunt versus the Baerveldt shunt for refractory glaucoma II: longer-term outcomes from a single surgeon. Ophthalmology. 2006 Jun;113(6):913-7. doi: 10.1016/j.ophtha.2006.02.029. PMID 16751034
- [Background] Goulet RJ 3rd, Phan AD, Cantor LB, WuDunn D. Efficacy of the Ahmed S2 glaucoma valve compared with the Baerveldt 250-mm2 glaucoma implant. Ophthalmology. 2008 Jul;115(7):1141-7. doi: 10.1016/j.ophtha.2007.10.034. Epub 2007 Dec 27. PMID 18164068
- [Background] Coleman AL, Hill R, Wilson MR, Choplin N, Kotas-Neumann R, Tam M, Bacharach J, Panek WC. Initial clinical experience with the Ahmed Glaucoma Valve implant. Am J Ophthalmol. 1995 Jul;120(1):23-31. doi: 10.1016/s0002-9394(14)73755-9. PMID 7611326
- [Background] Huang MC, Netland PA, Coleman AL, Siegner SW, Moster MR, Hill RA. Intermediate-term clinical experience with the Ahmed Glaucoma Valve implant. Am J Ophthalmol. 1999 Jan;127(1):27-33. doi: 10.1016/s0002-9394(98)00394-8. PMID 9932995
- [Background] Krishna R, Godfrey DG, Budenz DL, Escalona-Camaano E, Gedde SJ, Greenfield DS, Feuer W, Scott IU. Intermediate-term outcomes of 350-mm(2) Baerveldt glaucoma implants. Ophthalmology. 2001 Mar;108(3):621-6. doi: 10.1016/s0161-6420(00)00537-6. PMID 11237919
- [Background] Lloyd MA, Baerveldt G, Fellenbaum PS, Sidoti PA, Minckler DS, Martone JF, LaBree L, Heuer DK. Intermediate-term results of a randomized clinical trial of the 350- versus the 500-mm2 Baerveldt implant. Ophthalmology. 1994 Aug;101(8):1456-63; discussion 1463-4. doi: 10.1016/s0161-6420(94)31152-3. PMID 8058290
- [Background] Britt MT, LaBree LD, Lloyd MA, Minckler DS, Heuer DK, Baerveldt G, Varma R. Randomized clinical trial of the 350-mm2 versus the 500-mm2 Baerveldt implant: longer term results: is bigger better? Ophthalmology. 1999 Dec;106(12):2312-8. doi: 10.1016/S0161-6420(99)90532-8. PMID 10599663
- [Background] Nouri-Mahdavi K, Caprioli J. Evaluation of the hypertensive phase after insertion of the Ahmed Glaucoma Valve. Am J Ophthalmol. 2003 Dec;136(6):1001-8. doi: 10.1016/s0002-9394(03)00630-5. PMID 14644209
- [Background] Law SK, Nguyen A, Coleman AL, Caprioli J. Comparison of safety and efficacy between silicone and polypropylene Ahmed glaucoma valves in refractory glaucoma. Ophthalmology. 2005 Sep;112(9):1514-20. doi: 10.1016/j.ophtha.2005.04.012. PMID 16005977
- [Background] Ayyala RS, Harman LE, Michelini-Norris B, Ondrovic LE, Haller E, Margo CE, Stevens SX. Comparison of different biomaterials for glaucoma drainage devices. Arch Ophthalmol. 1999 Feb;117(2):233-6. doi: 10.1001/archopht.117.2.233. PMID 10037569
- [Background] Ayyala RS, Michelini-Norris B, Flores A, Haller E, Margo CE. Comparison of different biomaterials for glaucoma drainage devices: part 2. Arch Ophthalmol. 2000 Aug;118(8):1081-4. doi: 10.1001/archopht.118.8.1081. PMID 10922202
- [Background] Gedde SJ, Schiffman JC, Feuer WJ, Parrish RK 2nd, Heuer DK, Brandt JD; Tube Versus Trabeculectomy Study Group. The tube versus trabeculectomy study: design and baseline characteristics of study patients. Am J Ophthalmol. 2005 Aug;140(2):275-87. doi: 10.1016/j.ajo.2005.03.031. PMID 16086949
- [Background] Gedde SJ, Herndon LW, Brandt JD, Budenz DL, Feuer WJ, Schiffman JC. Surgical complications in the Tube Versus Trabeculectomy Study during the first year of follow-up. Am J Ophthalmol. 2007 Jan;143(1):23-31. doi: 10.1016/j.ajo.2006.07.022. Epub 2006 Sep 1. PMID 17054896
- [Background] Gedde SJ, Schiffman JC, Feuer WJ, Herndon LW, Brandt JD, Budenz DL. Treatment outcomes in the tube versus trabeculectomy study after one year of follow-up. Am J Ophthalmol. 2007 Jan;143(1):9-22. doi: 10.1016/j.ajo.2006.07.020. Epub 2006 Sep 1. PMID 17083910
- [Result] Christakis PG, Tsai JC, Zurakowski D, Kalenak JW, Cantor LB, Ahmed II. The Ahmed Versus Baerveldt study: design, baseline patient characteristics, and intraoperative complications. Ophthalmology. 2011 Nov;118(11):2172-9. doi: 10.1016/j.ophtha.2011.05.003. Epub 2011 Sep 9. PMID 21906813
- [Result] Christakis PG, Kalenak JW, Zurakowski D, Tsai JC, Kammer JA, Harasymowycz PJ, Ahmed II. The Ahmed Versus Baerveldt study: one-year treatment outcomes. Ophthalmology. 2011 Nov;118(11):2180-9. doi: 10.1016/j.ophtha.2011.05.004. Epub 2011 Sep 1. PMID 21889801
- [Result] Christakis PG, Tsai JC, Kalenak JW, Zurakowski D, Cantor LB, Kammer JA, Ahmed II. The Ahmed versus Baerveldt study: three-year treatment outcomes. Ophthalmology. 2013 Nov;120(11):2232-40. doi: 10.1016/j.ophtha.2013.04.018. Epub 2013 Jun 21. PMID 23796764
- [Result] Christakis PG, Kalenak JW, Tsai JC, Zurakowski D, Kammer JA, Harasymowycz PJ, Mura JJ, Cantor LB, Ahmed II. The Ahmed Versus Baerveldt Study: Five-Year Treatment Outcomes. Ophthalmology. 2016 Oct;123(10):2093-102. doi: 10.1016/j.ophtha.2016.06.035. Epub 2016 Aug 17. PMID 27544023

RESULTS

PARTICIPANT FLOW:
Groups:
- Ahmed Group: Ahmed FP7 Valve Implant
- Baerveldt Group: Baerveldt-350 Implant
Period: Overall Study
Arm/Group | Ahmed Group | Baerveldt Group
Started | 124 | 114
Completed | 89 | 82
Not Completed | 35 | 32
Not completed — Death | 8 | 12
Not completed — Lost to Follow-up | 27 | 20

BASELINE CHARACTERISTICS:
Groups:
- Ahmed Group: Patients received an Ahmed-FP7 valve implant at the time of surgery.
- Baerveldt Group: Patients received a Baerveldt-350 implant at the time of surgery.
- Total: Total of all reporting groups
Arm/Group | Ahmed Group | Baerveldt Group | Total
Number analyzed (Participants) | 124 | 114 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (17) | 67 (15) | 66 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 73 | 132
  Male | 65 | 41 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 15 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 13 | 28
  White | 96 | 86 | 182
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Intraocular Pressure [Mean (Standard Deviation); unit: mmHg] | 31.1 (10.5) | 31.7 (11.1) | 31.4 (10.8)
Glaucoma Medication Use [Mean (Standard Deviation); unit: medications] | 3.1 (1.0) | 3.1 (1.1) | 3.1 (1.0)
Prior Laser Therapies [Mean (Standard Deviation); unit: laser procedures] | 0.8 (1.1) | 1.0 (1.1) | 0.9 (1.1)
Prior Ocular Surgeries [Mean (Standard Deviation); unit: Ocular Surgeries] | 1.8 (1.3) | 1.6 (1.1) | 1.7 (1.2)
Mean logMAR (converted) Visual Acuity [Mean (Standard Deviation); unit: units on a scale] — LogMAR Visual Acuity is calculated by taking the log(Snellen Acuity/20). Normal vision (20/20) corresponds to 0 and complete blindness (no light perception, designated as 20/64000) corresponds to 3.5.
  Hence, the lower the logMAR value, the better the vision.
  units on a scale | 1.3 (1.0) | 1.3 (1.1) | 1.3 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Failure (Composite Measure)
Description: 1. IOP out of target range (5-18 mmHg inclusive) or <20% reduction from baseline for 2 consecutive visits after 3 months.
  2. De novo glaucoma surgery required (e.g., cyclodestructive procedure, additional tube shunt).
  3. Removal of the implant.
  4. Severe vision loss related to the surgery (endophthalmitis, suprachoroidal hemorrhage with vision loss, enucleation, evisceration, or phthisis bulbi) or progression to no light perception for any reason.
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Ahmed Group | Baerveldt Group
Number analyzed (Participants) | 124 | 114
participants | 63 | 40

2. Secondary Outcome: Intraocular Pressure (IOP)
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Ahmed Group: 124 patients were randomized to the Ahmed Group.
- Baerveldt Group: 114 patients were randomized to the Ahmed Group.
Arm/Group | Ahmed Group | Baerveldt Group
Number analyzed (Participants) | 124 | 114
mmHg | 16.6 (5.9) | 13.6 (5.0)

3. Secondary Outcome: Anti-glaucoma Medications
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: glaucoma medications
Arm/Group | Ahmed Group | Baerveldt Group
Number analyzed (Participants) | 124 | 114
glaucoma medications | 1.8 (1.5) | 1.2 (1.3)

4. Secondary Outcome: LogMAR Snellen Visual Acuity
Description: Visual acuity (VA) was tested monocularly (one eye at a time) using the manifest refraction adjusted for optical infinity using a standard Snellen Visual Acuity chart at 20 feet. Normal vision, or 20/20 vision, means that the participant can see at 20 feet what a healthy control can also see at 20 feet. Legal blindness, or 20/200 vision, means the participant can see at 20 feet what a healthy control can see at 200 feet. Hence, an increasing denominator implies visual impairment. Counting fingers was designated as 20/2000 vision, hand motions was 20/16000, light perception was 20/32000 and no light perception was 20/64000. To allow for appropriate statistical analysis, logMAR Snellen Visual Acuity was calculated using the formula: -logMAR (Snellen Acuity). This means that normal vision (20/20) would correspond to a value of 0, legal blindness (20/200) would correspond to a value of 1, and no light perception (20/64000) would correspond to 3.5.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: logMAR units on a scale
Arm/Group | Ahmed Group | Baerveldt Group
Number analyzed (Participants) | 124 | 114
logMAR units on a scale | 1.6 (1.0) | 1.6 (1.2)

5. Secondary Outcome: Number of Participants With Complications During or After Surgery
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ahmed Group | Baerveldt Group
Number analyzed (Participants) | 124 | 114
Participants | 78 | 79

6. Secondary Outcome: Number of Participants With Interventions After Surgery
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ahmed Group | Baerveldt Group
Number analyzed (Participants) | 124 | 114
Participants | 64 | 58

ADVERSE EVENTS:
Arm/Group | Ahmed Group | Baerveldt Group
Serious Adverse Events (participants affected / at risk) | 14/124 | 19/114
Other Adverse Events (participants affected / at risk) | 78/124 | 79/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ahmed Group (N=124) | Baerveldt Group (N=114)
Suprachoroidal Hemorrhage (Eye disorders) | 2 (2) | 3 (3)
Phthisis Bulbi (Eye disorders) | 1 (1) | 2 (2)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0)
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0)
Progression to no light perception (Eye disorders) | 7 (7) | 7 (7)
Device Explantation (Eye disorders) | 1 (1) | 2 (2)
Evisceration or enucleation (Eye disorders) | 3 (3) | 0 (0)
Hypotony Requiring Additional Surgery (Eye disorders) | 1 (1) | 6 (6)
Aqueous misdirection (Eye disorders) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ahmed Group (N=124) | Baerveldt Group (N=114)
Shallow Anterior Chamber (Eye disorders) | 18 (18) | 19 (19)
Choroidal Effusions (Eye disorders) | 16 (16) | 18 (18)
Tube Complications (Eye disorders) | 17 (17) | 19 (19)
Corneal Edema (Eye disorders) | 14 (14) | 14 (14)
Iritis (Eye disorders) | 9 (9) | 14 (14)
Cataract Progression (Eye disorders) | 11/34 (11) | 13/32 (13)
Encapsulated Bleb (Eye disorders) | 14 (14) | 4 (4)
Hyphema (Eye disorders) | 4 (4) | 6 (6)
Motility Disorder (Eye disorders) | 6 (6) | 2 (2)
High IOP requiring surgery (Eye disorders) | 19 (19) | 11 (11)
Other (Eye disorders) | 6 (6) | 7 (7)

LIMITATIONS AND CAVEATS:
1. Using predetermined IOP cutoffs may not reflect individual patient outcomes.
2. Visual field progression was not an outcome criteria due to the poor baseline vision of patients.
3. Results can only be applied to patients with advanced glaucoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No